CLINICAL TRIAL: NCT03501459
Title: Lymphocyte Markers As Predictors Of Responsiveness To Rituximab Among Patients With Idiopathic Nephrotic Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Isaac Liu, Professor Yap Hui Kim, National University Health System, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRC/NIG/0026/2008
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
The purpose of this study is to investigate if lymphocyte markers predict response to rituximab among patients with idiopathic nephrotic syndrome

ELIGIBILITY:
Inclusion Criteria:

* Age 1-18 years old at the time of diagnosis of nephrotic syndrome
* Steroid-dependent (SDNS) or steroid-resistant nephrotic syndrome (SDNS)

Exclusion Criteria:

* eGFR <60 ml/min per 1.73m2
* infantile onset of nephrotic syndrome
* nephrotic syndrome secondary to chronic infections such as hepatitis B, hepatitis C or human immunodeficiency virus, systemic lupus erythematosus, Henoch-Schönlein purpura, IgA nephropathy, membranoproliferative glomerulonephritis or membranous nephropathy
* current or previous therapy for tuberculosis
* presence of mutations in WT1, NPHS1, NPHS2 and TRPC6.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Response | 3 months
  Resolution of proteinuria (urine protein:creatinine <0.02 g/mmol or urine protein excretion <0.3 g/1.73m2/day) and ability to wean off prednisolone and calcineurin inhibitor at three months after the last dose of rituximab.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore